CLINICAL TRIAL: NCT02743910
Title: Plasma Tumor DNA and Pathologic Complete Response in Early-Stage, High-Risk Breast Cancer
Brief Title: Monitoring Plasma Tumor DNA in Early-Stage Breast Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Translational Breast Cancer Research Consortium (Other)
Responsible Party: Sponsor
Other Study IDs: TBCRC040; TBCRC 040 (Other: Translational Breast Cancer Research Consortium (TBCRC)); IRB00093688 (Other: JHMIRB)
Record Dates: First submitted 2016-04-15; First posted 2016-04-19 (Estimated); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
Keywords: preoperative; neoadjuvant; plasma tumor DNA; ptDNA
MeSH Terms: conditions — Breast Neoplasms | interventions — Blood Specimen Collection; Histocompatibility Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and tissue samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Stage II-III breast cancer: Up to 229 newly diagnosed stage II-III invasive HER2-positive or triple-negative breast cancer patients planning neoadjuvant therapy (NAT) will be enrolled. ptDNA blood samples as well as a representative tumor tissue sample from both the diagnostic and surgical procedure (if available) will be collected.
  Interventions: Other: ptDNA; Other: Tissue sample

INTERVENTIONS:
Other: ptDNA — Pre-operative blood samples for ptDNA will be collected at the time of diagnosis/prior to NAT, post-cycle 1/pre-cycle 2 of NAT, after all NAT/immediately before surgery, and post-operatively at 6, 12, 24, and 36 months, and annually thereafter if funding allows.
  Other Names: Blood sample
Other: Tissue sample — Representative tissue sample will be collected from the diagnostic biopsy (in all participants) and definitive surgery (if available)

SUMMARY:
This study is being done to see if it is possible to use blood samples to predict response to treatment in breast cancer patients receiving preoperative (or neoadjuvant) therapy. Research has shown that most breast cancers release tumor-specific DNA into the blood (that is, DNA that is specific to the tumor cells or cancer). This DNA can be detected in blood testing known as plasma tumor-DNA or "ptDNA." This DNA is separate from that found in the blood and tissue samples which serve as the "instruction book" or "genetic code" for the cells that make-up the human body. The changes in ptDNA before and after treatment, as well as after surgery, may also help investigators to understand more about a patient's risk of cancer returning and long-term outcomes.

DETAILED DESCRIPTION:
This is a prospectively designed study. Up to 229 newly diagnosed invasive HER2-positive or triple-negative breast cancer patients planning neoadjuvant therapy (NAT) will be enrolled. Blood samples will be collected pre-operatively at the time of diagnosis/prior to NAT, post-cycle 1/pre-cycle 2 of NAT, after all NAT/immediately before surgery, and post-operatively at 6, 12, 24, and 36 months, and annually thereafter if funding allows. Researchers will also collect representative tissue samples from the diagnostic biopsy (in all participants) and definitive surgery (if available). Additionally, to look at feasibility of tumor DNA analyses in urine samples, urine samples will be collected along with blood samples (urine tumor DNA or utDNA).

Next generation sequencing will be performed on core biopsies of all enrolled patients for tumor-specific mutations (TSM) discovery. Based on those findings, droplet digital PCR (ddPCR) on plasma DNA samples will also be performed to confirm the presence of the TSM in the plasma on diagnosis, and one TSM will be chosen to track as the plasma tumor DNA (ptDNA) mutation of interest. Investigators will perform ddPCR on pre-operative plasma DNA samples and will assess for the presence of ptDNA. Pathologists will assess surgical specimens for pathologic response (such as complete response/pCR and residual cancer burden/RCB). As primary endpoint, investigators will assess the number of patients with and without preoperative ptDNA who have pCR versus residual disease. As exploratory endpoints, the following will also be performed: (a) quantitative multiplex methylation-specific PCR (QM-MSP) in diagnostic biopsy and definitive residual surgery specimen; and, (b) the circulating methylated tumor DNA (cMethDNA) assay in plasma specimens (baseline and after NAT), and evaluate associations with pathologic response.

Additional endpoints include the association between plasma and tissue markers at baseline, after NAT, and (if available) during surveillance with long-term prognosis (invasive disease-free survival/IDFS and distant disease-free survival/DDFS).

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, histologically confirmed invasive breast cancer that is triple negative (estrogen receptor [ER], progesterone receptor [PR], and HER2-neu negative) or HER2-positive (any ER/PR status)
* Unresected, untreated breast cancer that is T2, T3, or T4a-c; any N (nodal status); and M0 (not metastatic)
* ECOG Performance Status of 0 or 1
* Planning to receive a neoadjuvant chemotherapy regimen containing a taxane ± an anthracycline for at least 4 cycles. Patients with HER2-positive disease must also be planning to receive HER2-targeted therapy.
* Diagnostic tumor material must be available for correlative analyses
* Patients must have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* No prior treatment for the current breast cancer, though prior use of selective estrogen receptor modulators (SERMs) or aromatase inhibitors (AIs) for the prevention of breast cancer is acceptable.
* Women who are pregnant or nursing are excluded.
* No history of another primary malignancy in the last 5 years prior to registration. Patients with prior history of in situ cancer or basal or localized squamous cell skin cancer are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed invasive HER2-positive or triple-negative breast cancer patients planning neoadjuvant therapy (NAT)
Sampling Method: Non-Probability Sample
Enrollment: 229 (Actual)
Dates: Start 2016-07; Primary Completion 2019-02 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Correlation of absence of plasma tumor DNA (ptDNA) with pathologic complete response (pCR) | 6 months
  To estimate the negative predictive value (NPV) of the absence of plasma tumor DNA (ptDNA) Tumor Specific Mutations (TSMs) after neoadjuvant therapy (NAT) for the absence of residual disease as defined by pathologic complete response (pCR) in stage II-III HER2-positive or triple negative breast cancer (TNBC)
  NPV = True Negative/True Negative + False Negative (probability that the disease is not present when the test is negative)

SECONDARY OUTCOMES:
Prognostic value of ptDNA for invasive disease-free survival and distant disease-free survival | 5 years
  To estimate the prognostic value of ptDNA for 5-year invasive disease-free survival (IDFS) and distant disease-free survival (DDFS) in TNBC patients following completion of loco-regional and systemic therapy
Correlation of absence of ptDNA with residual cancer burden (RCB) | 6 months
  To estimate the NPV of the absence of ptDNA TSMs after NAT for the absence of residual disease as defined by residual cancer burden (RCB) 0 or 1

CONTACTS AND LOCATIONS:
Overall Officials: Antonio C Wolff, M.D., Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No